CLINICAL TRIAL: NCT01048437
Title: Educating Missouri Patients About Preemptive Living Donor Transplantation: A Randomized Controlled Trial
Brief Title: Educating Missouri Patients About Preemptive Living Donor Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Missouri Kidney Program (Unknown); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy Waterman, PhD, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 080726
Record Dates: First submitted 2009-07-20; First posted 2010-01-13 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard transplant education (No Intervention): Missouri Kidney Program's standard Patient Education Program (PEP) transplant module.
- Transplant education with video (Experimental): Explore Transplant transplant module featuring video
  Interventions: Behavioral: Transplant education with video
- Transplant education with speakers (Experimental): Explore Transplant transplant module featuring live guest speakers.
  Interventions: Behavioral: Transplant education with speakers

INTERVENTIONS:
Behavioral: Transplant education with video — 1 hour standard transplant module is replaced with the Explore Transplant presentation and 20 minute video featuring transplant patients and donors
  Arms: Transplant education with video
Behavioral: Transplant education with speakers — 1 hour standard transplant module is replaced with the Explore Transplant presentation and 3 live speakers: 1 deceased donor recipient, 1 living donor recipient and 1 living donor
  Arms: Transplant education with speakers

SUMMARY:
This study is a group-randomized controlled trial to explore whether improved community transplant education for renal patients not yet on dialysis could increase patients' willingness to pursue preemptive living donor transplant (PLDT) and PLDT rates.

DETAILED DESCRIPTION:
Preemptive living donor transplant (PLDT), where renal patients get a living donor transplant before their kidneys fail, has better graft survival and lower mortality rates than living donor transplant following dialysis. However, not all renal patients and their living donors know about or consider living donation before a patient starts dialysis; To date, patients and donors presenting for PLDT are more likely to be Caucasian, of higher socioeconomic status, and more knowledgeable about transplant. To reach all patients newly diagnosed with kidney disease, the Missouri Kidney Program conducts a community Patient Education Program (PEP) outlining patients' transplant and dialysis options. Since 1994, approximately 2000 Missouri patients newly diagnosed with kidney disease and their family members have attended 2-day PEP classes. However, the current PEP transplant module does not significantly increase patients' willingness to pursue PLDT. Through a previous HRSA grant, Dr. Waterman designed the "Explore Transplant" education program based on Prochaska's Transtheoretical Model of Behavioral Change and her previous research to address key gaps in patients' living donation knowledge and to motivate patients to consider living donation. If funded, this study would conduct a group-randomized controlled trial to explore whether improved community transplant education for renal patients not yet on dialysis could increase patients' willingness to pursue PLDT and PLDT rates. Secondary objectives of the study are: (2) to increase rural and minority patients' access to transplant education, and (3) to describe racial, social, economic, and other influences affecting patients' PLDT willingness. The study design is a group-randomized controlled trial of 300 patients in 30 PEP classes in St. Louis, Springfield, and Kansas City, MO; patients and their family members in 15 classes will be randomized to receive the "Explore Transplant" education module, while 15 control classes will receive the traditional PEP transplant education. Across the education and control PEP classes we will compare: (1) increased willingness to pursue PLDT using baseline and follow-up attitudinal patient surveys, and (2) rates of living donation by tracking whether patients and their living donors present to any Missouri transplant center. At the conclusion of the study, we will have learned important information about how to reach and educate patients who have not yet begun dialysis and have developed a PLDT program that could be utilized in physicians' offices and by other organizations serving renal patients to increase living donation rates.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Attend all 6 education modules
* 18+ years of age
* Have given consent by signing informed consent
* Speak and understand English
* Can read and understand questionnaires

Exclusion Criteria:

* Patients who do not speak and understand English (material is presented orally)
* Patients who cannot read and understand the questionnaires
* Patients who are 17 years of age or younger

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Willingness to pursue preemptive living donor transplant | pre and post-class

SECONDARY OUTCOMES:
Preemptive living donor transplant rates | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Waterman, PhD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Missouri Kidney Program, Overland Park, Kansas
  - Missouri Kidney Program, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - Missouri Kidney Program, St Louis, Missouri
  - Missouri Kidney Program, Warrensburg, Missouri